CLINICAL TRIAL: NCT00113074
Title: Blood Pressure Control in Hypertensive Smokers
Brief Title: Preventing Weight Gain and Controlling Blood Pressure During Smoking Cessation in Hypertensive Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark Vander Weg (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Mark Vander Weg, Mark W. Vander Weg, PhD, University of Iowa, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 200611724; R01HL072782 (NIH)
Record Dates: First submitted 2005-06-03; First posted 2005-06-06 (Estimated); Results first posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension | interventions — Nicotine Replacement Therapy; Diet

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Weight management and blood pressure control intervention
  Interventions: Drug: Nicotine Replacement Therapy; Behavioral: Diet
- 3 (Active Comparator): Self-help materials targeting lifestyle modification
  Interventions: Drug: Nicotine Replacement Therapy; Behavioral: Diet
- 2 (Experimental): Weight management intervention
  Interventions: Drug: Nicotine Replacement Therapy; Behavioral: Diet

INTERVENTIONS:
Drug: Nicotine Replacement Therapy — Nicotine replacement therapy program
Behavioral: Diet — Diet program

SUMMARY:
The purpose of this study is to develop effective interventions that assist individuals with high blood pressure to quit smoking and prevent weight gain.

DETAILED DESCRIPTION:
BACKGROUND:

High blood pressure (BP), or hypertension, is a major risk factor for cardiovascular morbidity and mortality. Hypertension is associated with an elevated risk for several cardiovascular complications, including coronary heart disease, peripheral vascular disease, congestive heart failure, and stroke, as well as an increased risk for renal disease. Although there have been significant advances in the detection and treatment of high BP, approximately one in four adults in the United States is hypertensive. Cigarette smoking accounts for more than 400,000 premature deaths each year in this country alone, making it the leading cause of morbidity and mortality. Evidence from several epidemiological studies has demonstrated that, at any level of BP, smoking substantially increases the risk for all cardiovascular complications associated with hypertension. While cigarette smoking and hypertension both increase the risk of cardiovascular disease, these two risk factors act synergistically to produce a greater risk than their combined independent effects. Despite the considerable health risks, smoking among people with hypertension is very common, with a prevalence approaching that observed among those with normal BP. Unfortunately, although quitting smoking is especially important for patients with high BP, smoking cessation produces a nontrivial weight gain, averaging 5 kg, which may exacerbate hypertension in many patients with the disorder. Several studies have documented significant elevations in BP following smoking cessation, as well as increases in the prevalence of hypertension after quitting smoking. As such, it is important to develop effective interventions that assist in quitting smoking and preventing weight gain.

DESIGN NARRATIVE:

The objective of the trial is to recruit 750 smokers with Stage 1 hypertension or prehypertension (based on JNC VII criteria). The trial will provide all participants with a brief, validated, combined behavioral and pharmacologic smoking cessation intervention. Additionally, the study will randomly assign participants who are abstinent from smoking upon completing the cessation intervention to either a 12-week weight management and BP control program or self-help materials targeting lifestyle modification. The primary endpoint is change in BP among quit smokers at a one-year follow-up. Secondary endpoints include changes in body weight, dietary intake, urinary sodium excretion, physical activity, and relapse to smoking. Exploratory endpoints include changes in hypertensive status (e.g., movement from prehypertensive to hypertensive by JNC VII criteria) and changes in BP medication status. This is a multi-site clinical trial, with study locations in Rochester, Minnesota, and Iowa City, IA. The Rochester, MN site is currently closed for recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Smoke at least 5 cigarettes/day (or have quit within the last 6 weeks to enter the study for the weight gain prevention and BP control interventions)
* Pre-hypertensive or Stage I hypertension (systolic BP from 120 to 159 and/or diastolic BP from 80 to 99 mm Hg). Antihypertensive medications are not criteria for exclusion provided that BP is not over 160/100 mm Hg)
* Access to a telephone

Exclusion Criteria:

* History of unstable cardiovascular disease, including myocardial infarction, stroke, and unstable angina within three months of study start
* Coronary artery bypass grafting or angioplasty/stent within three months of study start
* Cardiac dysrhythmia treated with anti-arrhythmia medication, except stable atrial fibrillation
* Untreated hyperthyroidism or pheochromocytoma
* History of congestive heart failure (NYHA Class III or IV)
* ECG evidence of 2nd or 3rd degree atrioventricular block
* Uncontrolled or Stage II Hypertension as defined as BP consistently above 160/100 mm Hg
* History of severe liver or kidney failure
* Current substance abuse (includes alcohol use in excess of 21 drinks a week)
* Presence of an unstable psychiatric condition
* Severe chronic obstructive pulmonary disease
* Symptomatic peripheral vascular disease
* Pulmonary hypertension with shortness of breath
* Congenital or valvular heart disease with shortness of breath
* Current use of a medication that may interfere with primary study endpoints or that may increase the risk of side effects from study medication that cannot be discontinued
* Pregnant or plans to become pregnant within the next year
* Planning to move out of the area or travel extensively during the intervention
* Any medical condition that would preclude any additional changes in diet
* Unable to further modify physical activity routine
* Cannot engage in moderate intensity exercise (e.g., walking)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2004-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark W. Vander Weg, PhD, Principal Investigator — University of Iowa, Carver College of Medicine, Department of Internal Medicine
Locations (2):
- United States (2):
  - University of Iowa, Carver College of Medicine, Department of Internal Medicine, Division of General Internal Medicine, Iowa City, Iowa
  - Mayo Clinic College of Medicine, Rochester, Minnesota

REFERENCES:
- [Background] Vander Weg MW, Klesges RC, Ebbert JO, Lichty EJ, DeBon M, North F, Schroeder DR, Dubbert PM. Trial design: blood pressure control and weight gain prevention in prehypertensive and hypertensive smokers: the treatment and prevention study. Contemp Clin Trials. 2008 Mar;29(2):281-92. doi: 10.1016/j.cct.2007.07.003. Epub 2007 Jul 19. PMID 17716953

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 - Weight Management and Blood Pressure Control Intervention: Weight management and blood pressure control intervention
  Nicotine Replacement Therapy: Nicotine replacement therapy program
  Diet: Diet program
- 3 - Self-help Materials Targeting Lifestyle Modification: Self-help materials targeting lifestyle modification
  Nicotine Replacement Therapy: Nicotine replacement therapy program
  Diet: Diet program
- 2 - Weight Management Intervention: Weight management intervention
  Nicotine Replacement Therapy: Nicotine replacement therapy program
  Diet: Diet program
Period: Overall Study
Arm/Group | 1 - Weight Management and Blood Pressure Control Intervention | 3 - Self-help Materials Targeting Lifestyle Modification | 2 - Weight Management Intervention
Started | 49 | 43 | 47
Completed | 39 | 33 | 33
Not Completed | 10 | 10 | 14
Not completed — Lost to Follow-up | 10 | 10 | 14

BASELINE CHARACTERISTICS:
Population: Based on participants who successfully quit smoking during Phase I of the study and were subsequently randomized to treatment conditions
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 - Weight Management and Blood Pressure Control Intervention | 3 - Self-help Materials Targeting Lifestyle Modification | 2 - Weight Management Intervention | Total
Number analyzed (Participants) | 49 | 43 | 47 | 139
Age, Categorical [Count of Participants; unit: Participants] — Population: One participant had missing data on this variable.
  Participants
    number analyzed (Participants) | 49 | 43 | 46 | 138
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 45 | 38 | 41 | 124
    >=65 years | 4 | 5 | 5 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (13.8) | 46.6 (13.1) | 47.3 (14.2) | 46.6 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant had missing data on this variable.
  Participants
    number analyzed (Participants) | 49 | 43 | 46 | 138
    Female | 19 | 13 | 18 | 50
    Male | 30 | 30 | 28 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant had missing data on this variable.
  Participants
    number analyzed (Participants) | 49 | 43 | 46 | 138
    Hispanic or Latino | 2 | 2 | 0 | 4
    Not Hispanic or Latino | 47 | 41 | 46 | 134
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant had missing data on this variable.
  Participants
    number analyzed (Participants) | 49 | 43 | 46 | 138
    American Indian or Alaska Native | 1 | 0 | 1 | 2
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 3 | 3 | 0 | 6
    White | 44 | 39 | 45 | 128
    More than one race | 1 | 1 | 0 | 2
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 49 | 43 | 47 | 139
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Data missing for 5 participants
  mmHg
    number analyzed (Participants) | 48 | 42 | 43 | 133
    (all) | 130.3 (11.3) | 131.6 (11.5) | 128.8 (12.2) | 130.2 (11.6)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Data missing for 5 participants.
  mmHg
    number analyzed (Participants) | 48 | 42 | 43 | 133
    (all) | 79.3 (8.4) | 79.1 (8.7) | 77.9 (9.5) | 78.8 (8.8)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Data missing for three participants
  kg/m^2
    number analyzed (Participants) | 48 | 43 | 44 | 135
    (all) | 30.6 (7.6) | 29.5 (6.2) | 30.0 (6.1) | 30.1 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure at One Year Among People Who Have Quit Smoking
Description: Change in systolic blood pressure in mmHg
Time Frame: Measured at Year 1
Population: Participants still abstinent from smoking at one year who attended 12-month follow-up.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Groups:
- Weight Management and Blood Pressure Control Intervention: Weight management and blood pressure control intervention
  Nicotine Replacement Therapy: Nicotine replacement therapy program
  Diet: Diet program
- Self-help Materials Targeting Lifestyle Modification: Self-help materials targeting lifestyle modification
  Nicotine Replacement Therapy: Nicotine replacement therapy program
  Diet: Diet program
- Weight Management Intervention: Weight management intervention
  Nicotine Replacement Therapy: Nicotine replacement therapy program
  Diet: Diet program
Arm/Group | Weight Management and Blood Pressure Control Intervention | Self-help Materials Targeting Lifestyle Modification | Weight Management Intervention
Number analyzed (Participants) | 23 | 12 | 14
millimeters of mercury (mmHg) | -1.78 (12.81) | -0.17 (11.42) | -1.64 (10.62)

2. Primary Outcome: Change in Diastolic Blood Pressure at One Year Among People Who Have Quit Smoking
Description: Change in diastolic blood pressure in mmHg
Time Frame: Measured at Year 1
Population: Participants still abstinent from smoking at one year who attended 12-month follow-up.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Weight Management and Blood Pressure Control Intervention | Self-help Materials Targeting Lifestyle Modification | Weight Management Intervention
Number analyzed (Participants) | 23 | 12 | 14
millimeters of mercury (mmHg) | -0.35 (8.62) | -1.17 (5.77) | 0.93 (7.38)

3. Secondary Outcome: Changes in Body Weight
Description: Change in body weight in pounds from randomization to 12 months.
Time Frame: Measured at Year 1
Population: Randomized participants who were still abstinent from smoking at 12 months and who provided weight data.
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Weight Management and Blood Pressure Control Intervention | Self-help Materials Targeting Lifestyle Modification | Weight Management Intervention
Number analyzed (Participants) | 24 | 12 | 15
Pounds | 3.07 (10.40) | 2.73 (9.17) | 6.20 (7.99)

4. Secondary Outcome: Dietary Intake - Fruit and Vegetable Consumption
Description: Change in self-reported daily fruit and vegetable consumption from randomization to 12 months. Fruit and vegetable consumption was measured by self-report using a dietary screener, which provides results in the form of number of servings per day.
Time Frame: Measured at Year 1
Population: Randomized participants who were still abstinent from tobacco use at 12 months and who provided follow-up data.
Measure: Mean (Standard Deviation); unit: Servings of fruits and vegetables/day
Arm/Group | Weight Management and Blood Pressure Control Intervention | Self-help Materials Targeting Lifestyle Modification | Weight Management Intervention
Number analyzed (Participants) | 23 | 12 | 15
Servings of fruits and vegetables/day | 1.32 (3.31) | -3.46 (6.49) | -0.29 (3.31)

5. Secondary Outcome: Urinary Sodium Chloride Excretion
Description: Percent change in urinary sodium chloride (NaCL) from randomization to one-year
Time Frame: Measured at Year 1
Population: Participants from Rochester site who were abstinent from smoking at one-year and who provided urinary chloride data at randomization visit and one-year. Urinary chloride data are not available from the Iowa City site.
Measure: Mean (Standard Deviation); unit: Percent change in urinary NaCL excretion
Groups:
- 1 - Weight Management and Blood Pressure Control Intervention: Weight management and blood pressure control intervention
  Nicotine Replacement Therapy: Nicotine replacement therapy program
  Diet: Diet program focused on energy restriction, sodium restriction, and DASH diet
- 3 - Self-help Materials Targeting Lifestyle Modification: Self-help materials targeting lifestyle modification
  Nicotine Replacement Therapy: Nicotine replacement therapy program
  Diet: Self-help diet intervention focused on weight management
- 2 - Weight Management Intervention: Weight management intervention
  Nicotine Replacement Therapy: Nicotine replacement therapy program
  Diet: Diet program focused on energy restriction
Arm/Group | 1 - Weight Management and Blood Pressure Control Intervention | 3 - Self-help Materials Targeting Lifestyle Modification | 2 - Weight Management Intervention
Number analyzed (Participants) | 3 | 6 | 7
Percent change in urinary NaCL excretion | .01 (.10) | .05 (.18) | -.05 (.07)

6. Secondary Outcome: Physical Activity: Leisure Time Physical Activity in METs
Description: Change in leisure time physical activity in metabolic equivalents (METs) from randomization to one-year. METs reflect the ratio of working metabolic rate relative to resting metabolic rate, and are expressed as the energy expended per unit of time. For this study, METs were measured based on self-reported physical activity using the International Physical Activity Questionnaire (IPAQ) and are reported in the form of MET minutes.
Time Frame: Measured at Year 1
Population: Participants who remained abstinent from tobacco use and who provided physical activity data at randomization and one-year.
Measure: Mean (Standard Deviation); unit: MET minutes
Arm/Group | Weight Management and Blood Pressure Control Intervention | Self-help Materials Targeting Lifestyle Modification | Weight Management Intervention
Number analyzed (Participants) | 21 | 10 | 14
MET minutes | 293.7 (1000.4) | 277.5 (1862.4) | -1383.5 (2557.6)

7. Secondary Outcome: Relapse to Smoking
Description: Number of participants who self-reported tobacco use during the last seven-days.
Time Frame: Measured at Year 1
Population: Participants randomized to treatment groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Weight Management and Blood Pressure Control Intervention | Self-help Materials Targeting Lifestyle Modification | Weight Management Intervention
Number analyzed (Participants) | 49 | 43 | 46
Participants | 24 | 30 | 30

8. Secondary Outcome: Dietary Intake - Dietary Fat Consumption
Description: Change in daily dietary fat consumption from randomization to 12 months.
Time Frame: Measured at Year 1
Population: Randomized participants who were still abstinent from tobacco use at 12 months and who provided follow-up data.
Measure: Mean (Standard Deviation); unit: Grams of dietary fat consumed/d
Arm/Group | Weight Management and Blood Pressure Control Intervention | Self-help Materials Targeting Lifestyle Modification | Weight Management Intervention
Number analyzed (Participants) | 21 | 12 | 14
Grams of dietary fat consumed/d | -2.39 (4.71) | -0.81 (2.99) | -0.88 (2.79)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Coded for intensity (Mild, Moderate, Severe, Unknown), Seriousness (Not serious, Serious/not life threatening, Life threatening, Fatal), Relationship to study (Not related, Remote, Possible, Probable, Definite), Action (None, Concomitant medication required, Study drug discontinued temporarily, Study drug discontinued permanently, MD visit, Hospitalization, Other, Unknown), Outcome (Resolved, Continues resolving, Continuing but stable, Worsening, Other, Unknown), dates, and duration.
Arm/Group | Weight Management and Blood Pressure Control Intervention | Self-help Materials Targeting Lifestyle Modification | Weight Management Intervention
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/43 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/49 | 1/43 | 1/47
Other Adverse Events (participants affected / at risk) | 24/49 | 19/43 | 24/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Management and Blood Pressure Control Intervention (N=49) | Self-help Materials Targeting Lifestyle Modification (N=43) | Weight Management Intervention (N=47)
Kidney Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — Kidney Cancer diagnosed in one participant and determined not to be related to study procedures.
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — One participant was diagnosed with prostate cancer. It was determined not to be related to study procedures.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Management and Blood Pressure Control Intervention (N=49) | Self-help Materials Targeting Lifestyle Modification (N=43) | Weight Management Intervention (N=47)
Itching/irritation/rash/pain at nicotine patch site (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6) | 6 (6)
Other musculoskeletal pain/injury (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 3 (3) — Miscellaneous musculoskeletal pain, injury, or disorders that were not captured in the categories of: 1) bone fracture, 2) back pain, soreness, or sprain, 3) or osteopenia or osteoporosis, each of which were assessed as separate categories.
Nightmares/strange or vivid dreams (Nervous system disorders) | 2 (2) | 2 (2) | 4 (4)
Upper respiratory infection/cold (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 10 (10) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT00113074/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT00113074/SAP_001.pdf
  • Informed Consent Form (2009-11-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT00113074/ICF_002.pdf